CLINICAL TRIAL: NCT01425424
Title: Prediabetes, Prehypertension and Vitamin D Supplementation - A Practice Based Clinical Intervention Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI was leaving Pennington
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Frank Greenway, Princiapal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PBRC 10036
Record Dates: First submitted 2011-08-10; First posted 2011-08-30 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Prediabetes; Prehypertension
Keywords: Vitamin D; Prediabetes; Prehypertension
MeSH Terms: conditions — Prediabetic State; Prehypertension | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fasting glucose (blood sugar) (Experimental): This group is associated with a diagnosis of prediabetes
  Interventions: Other: Vitamin D supplementation
- Resting Blood pressure (Experimental): This group is associated with a diagnosis of prehypertension.
  Interventions: Other: Vitamin D supplementation
- Fasting Glucose & Resting Blood Pressure (Experimental): coexisting prediabetes and prehypertension
  Interventions: Other: Vitamin D supplementation

INTERVENTIONS:
Other: Vitamin D supplementation — Vitamin D
  Other Names: Vitamin D

SUMMARY:
This randomized, double-blind, placebo-controlled, multi-site study is to reverse modest elevations of fasting blood sugar (prediabetes) and resting blood pressure(Prehypertension) or both co existing prediabetes and prehypertension by increasing blood levels of vitamin D. This may reduce the chances of developing diabetes or high blood pressure or both later in life.

DETAILED DESCRIPTION:
Study visits will measure temperature, fasting glucose, resting blood pressure, respiratory rate, height, weight and waist circumference. A brief medical History will be taken, followed by an abbreviated physical exam. A blood test to check your vitamin D level and routine chemistry including a complete lipid profile, liver and kidney function will be completed.

Based on your fasting glucose and/or resting blood pressure you will be in one of the three arms: prediabetes (arm 1), prehypertension (arm 2) or co-existing prediabetes and prehypertension (arm 3). After determining the arm of the study you are in, you will be randomly assigned to receive either a placebo or vitamin D supplementation.

If you are in the first arm with prediabetes (fasting glucose 100-125 mg/dL), the primary outcome measure will change in fasting glucose at 8 weeks, 16 weeks and every 3 months until you are in the study up to 5 years. If you are in the second arm with prehypertension (resting blood pressure 120-139/80-89 mm Hg), the primary outcome measure will change in resting blood pressure at 8 weeks, 16 weeks and every 3 months until you are in the study up to 5 years. If you are in third arm with prediabetes and prehypertension, both these measures will be taken at 8 weeks, 16 weeks and every 3 months until you are in the study up to 5 years. A repeat blood test to check vitamin D levels will be done at 8 and 16 weeks (and periodically as necessary) during the study.

Other measures will be taken as are routine in your doctor's office.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male or Female 18 years or older presenting to The America Family Practice, Physicians Care Center offices or Egan Wellness Clinic/Anti-Aging & Skin Care Spa.
* Agreeable to treatment with placebo or vitamin D 1000IU twice a day with food.

Exclusion Criteria:

* Women who are pregnant or nursing
* Anyone with chronic medical conditions requiring regular intake of any prescription medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Prediabetes, Prehypertension and Vitamin D supplementation- A practice based clinical intervention | 8 weeks
  An analysis of the fasting glucose, resting blood pressure and/or both will be performed. A blood test to check your vitamin D level and routine chemistry including a complete lipid profile, liver and kidney function will also be done. At the end of 8 weeks fasting blood glucose and resting blood pressure will be measured. If the desired results (fasting glucose less than 100 mg/dL and/or resting blood pressure less than 120/80 mm Hg) are not seen these measures will be repeated at 16 weeks. You will be asked to stay in the study for up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Alok Gupta, MD, AAFP, FASH, Principal Investigator — Pennington Biomedical Research Center
Locations (7):
- United States (7):
  - Physicians Care Center, Baton Rouge, Louisiana
  - Bradley L. Meek, MD, Internal Medicine at Hennessy, Baton Rouge, Louisiana
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Metabolic Clinic Women's Hospital, Baton Rouge, Louisiana
  - Egan Wellness Clinic/AntiAging & Skin Care Spa, Covington, Louisiana
  - Amarica Family Practice Office (Second Location), Durham, North Carolina
  - Amarica Family Practice Office (First Location), Roxboro, North Carolina